CLINICAL TRIAL: NCT04760821
Title: Prevention of Acute Myocardial Injury by Trimetazidine in Patients Hospitalized for Moderate to Severe Acute Respiratory Syndrome Caused by SARS-CoV-2
Brief Title: Prevention of Acute Myocardial Injury by Trimetazidine in Patients Hospitalized for COVID-19
Acronym: PREMIER
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ministry of Health, Brazil (Other Government)
Collaborators: InCor Heart Institute (Other)
Responsible Party: Principal Investigator, Luis Henrique W Gowdak, MD, PhD, Clinical Scientist, InCor Heart Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SDC5100/20/129
Record Dates: First submitted 2021-02-17; First posted 2021-02-18 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Acute Respiratory Distress Syndrome; Covid19; Myocardial Injury
Keywords: Acute Respiratory Distress Syndrome; Coronavirus; Myocardial Injury; Troponin; Trimetazidine
MeSH Terms: conditions — Respiratory Distress Syndrome; COVID-19; Coronavirus Infections | interventions — Trimetazidine

STUDY DESIGN:
Intervention Model Description: Patients admitted for moderate to severe acute respiratory distress syndrome caused by the SARS-CoV2 will be randomized to usual care or usual care + trimetazidine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Patients ascribed to the Usual Care group will receive the standard of care for the management of patients admitted with moderate to severe acute respiratory distress syndrome due to SARS-CoV2. Usual Care means the clinical protocol approved by the enrolling center.
- Trimetazidine (Experimental): Patients ascribed to the Usual Care group will receive the standard of care for the management of patients admitted with moderate to severe acute respiratory distress syndrome due to SARS-CoV2 plus trimetazidine.Usual Care means the clinical protocol approved by the enrolling center.
  Interventions: Drug: Trimetazidine

INTERVENTIONS:
Drug: Trimetazidine — Trimetazidine 35mg bid in patients with GFR above 60mL/min. Trimetazidine 35mg od in patients with GFR between 30 and 60mL/min.
  Arms: Trimetazidine

SUMMARY:
Acute myocardial injury has been a finding of variable frequency among patients diagnosed with COVID-19. It is now recognized that cTnI levels are strongly associated with increased mortality. The mechanisms underlying the myocardial injury remain unknown, and it is not clear whether they reflect local/systemic inflammatory process and/or cellular ischemia.

Both myocardial ischemia and ventricular dysfunction result in dramatic changes in mitochondrial oxidative metabolism. These changes involve an increase in the rate of cytoplasmic anaerobic glycolysis to compensate for the decrease in mitochondrial adenosine triphosphate (ATP) production. The rest of the mitochondrial oxidative metabolism originates mainly from the β-oxidation of free fatty acids, which occurs at the expense of glucose oxidation.

Trimetazidine is a competitive inhibitor of the enzyme 3-ketoacyl coenzyme A (CoA) long-chain thiolase (3-KAT), the last enzyme involved in the oxidation of fatty acids. Stimulation of glucose oxidation by trimetazidine results in a better coupling between glycolysis and glucose oxidation, with a consequent decrease in lactate production and intracellular acidosis, present in situations of myocardial ischemia or heart failure.

Thus, the PREMIER-COVID-19 study was designed to test the hypothesis that the use of trimetazidine associated with usual therapy in patients admitted with a diagnosis of moderate to severe acute respiratory syndrome by SARS-CoV2 infection reduces the extent of acute myocardial injury assessed by the peak release of ultra-sensitive troponin compared to usual therapy.

DETAILED DESCRIPTION:
Acute myocardial injury, defined by increased levels of high-sensitivity cardiac troponin I (cTnI), has been a finding of variable frequency among patients diagnosed with COVID-19. This myocardial impairment can occur in the form of acute myocarditis or an injury secondary to the imbalance between oxygen supply and demand (type 2 myocardial infarction). It is now recognized that cTnI levels are strongly associated with increased mortality. The mechanisms underlying the myocardial injury remain unknown, and it is not clear whether they reflect local/systemic inflammatory process and/or cellular ischemia.

Both myocardial ischemia and ventricular dysfunction result in dramatic changes in mitochondrial oxidative metabolism. These changes involve an increase in cytoplasmic anaerobic glycolysis rate to compensate for the decrease in mitochondrial ATP production. Unfortunately, the increase in glycolysis exceeds the subsequent mitochondrial oxidation capacity of pyruvate (glucose oxidation) derived from glycolysis, resulting in the intracellular accumulation of lactate and protons. The protons produced from this decoupling between glycolysis and glucose oxidation contribute to a rupture in ionic homeostasis and myocardial cells, resulting in lower cardiac efficiency. In both the ischemic heart and the insufficient heart, the rest of the mitochondrial oxidative metabolism originates mainly from the β-oxidation of free fatty acids, which occurs at the expense of glucose oxidation.

Trimetazidine is a competitive inhibitor of the enzyme 3-ketoacyl CoA long-chain thiolase (3-KAT), the last enzyme involved in the oxidation of fatty acids. Stimulation of glucose oxidation by trimetazidine results in a better coupling between glycolysis and glucose oxidation, with a consequent decrease in lactate production and intracellular acidosis present in situations of myocardial ischemia or heart failure.

Thus, the PREMIER-COVID-19 study (open and randomized) was designed to test the hypothesis that the use of trimetazidine associated with usual therapy in patients admitted with a diagnosis of moderate to severe acute respiratory syndrome by SARS-CoV2 infection reduces the extent of acute myocardial injury assessed by the peak release of ultra-sensitive troponin compared to usual therapy. Investigators will also assess, as secondary outcomes, the impact on clinical evolution to more severe forms (admission to the intensive care unit or the need for mechanical ventilatory support, length of stay in hospital and in-hospital mortality).

ELIGIBILITY:
A. Inclusion Criteria:

1. Clinical diagnosis of moderate to severe acute respiratory syndrome due to SARS-CoV2 defined as:

   1.1. Tachypnea: > 24 breaths per minute 1.2. Hypoxemia: arterial oxygen saturation <94% in room air by pulse oximetry 1.3. Presumptive (or confirmed) diagnosis of SARS-Cov2 infection by at least one of the following criteria:
   1. Polymerase chain reaction assay (+) for SARS-CoV2
   2. Serology (+) for SARS-CoV2
   3. SARS-CoV2 antigen diagnostic tests (+)
   4. Chest CT with findings suggestive of the diagnosis of COVID-19 in the presence of medical history or clinical signs compatible with the diagnosis of COVID-19
2. Signature of the Informed Consent Form

B. Exclusion Criteria:

1. Chronic renal dysfunction stage 4 (GFR <30mL / min / 1.73m2 calculated by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation
2. Patient on renal replacement therapy by dialysis
3. Pregnant and lactating women
4. Previous use of trimetazidine less than two weeks before hospital admission
5. Any clinical condition at the investigator´s discretion likely to be associated with elevation of baseline hs-troponin >99th percentile

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-12-10 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
High-sensitivity cardiac troponin | From enrollment until at least ten days (moderate cases) or twenty days (severe cases) after the beginning of symptoms AND 24 hours without fever AND with improvement in symptoms.
  Concentration levels of plasma high-sensitivity cardiac troponin

SECONDARY OUTCOMES:
All-cause mortality assessed at 30 days following randomization | From the first 30 days after randomization
  Percentage of patients who died from all causes during hospitalization
Admission in ICU assessed at 30 days following randomization | From the first 30 days after randomization
  Percentage of patients admitted to the Intensive Care Unit
Mechanical respiratory support assessed at 30 days following randomization | From the first 30 days after randomization
  Percentage of patients admitted to the Intensive Care Unit who needed mechanical respiratory support
ICU-free days assessed at 30 days following randomization | From the first 30 days after randomization
  Time (in days) out of the ICU
Hospital-free days assessed at 30 days following randomization | From the first 30 days after randomization
  Time (in days) out of the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Luis Henrique Wolff Gowdak, MD, PhD, Study Chair — InCor (HC-FMUSP); Felipe Gallego Lima, MD, Principal Investigator — InCor (HC-FMUSP)
Locations (1):
- Heart Institute (InCor-HCFMUSP), São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No